CLINICAL TRIAL: NCT04765683
Title: Video, Telephone or Face-to-face Surgical Consultations: a Survey of Patients' and Surgeons' Views
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Principal Investigator, Sebastian Aspinall, Consultant General Surgeon, Chief Investigator, University of Aberdeen
Other Study IDs: 287686
Record Dates: First submitted 2020-12-18; First posted 2021-02-21 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Surgery
Keywords: outpatient consultation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Attending surgical outpatients
  Interventions: Other: questionnaire
- Surgeons: Running surgical outpatients
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Survey of views on outpatient consultation format

SUMMARY:
This study will send out questionnaires to surgical outpatients and surgeons to gather their views on the appropriate type of surgical outpatient consultation in different clinical scenarios, in order to establish a guideline for surgical outpatient planning.

DETAILED DESCRIPTION:
As above - this study will send out questionnaires to surgical outpatients and surgeons to gather their views on the appropriate type of surgical outpatient consultation in different clinical scenarios, in order to establish a guideline for surgical outpatient planning.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS

Adults attending general surgical outpatients in Aberdeen Royal Infirmary during the study period presenting with:

* lumps and bumps
* hernias
* biliary problems
* jaundice
* abdominal pain/mass/weight loss
* gastro-oesophageal reflux
* dysphagia
* change in bowel habit
* anorectal problems
* thyroid nodules
* parathyroid disease
* adrenal masses

SURGEONS

Consultant General Surgeons in NHS Grampian / Tayside and Highlands

Exclusion Criteria:

PATIENTS

* lacking capacity
* without language skills to answer questionnaires or ability to understand questionnaires
* children < 16yrs (No upper age limit)
* patients presenting as emergencies
* patients unwilling to complete questionnaires.

SURGEONS

- trainee surgeons.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: General surgical outpatients General surgeons
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
appropriate type of surgical outcome | June 2021
  What type of surgical outpatient consultation is appropriate for different clinical scenarios i.e. new patient, review patient, post-operative results, breaking bad news, cancer follow-up? This will be assessed by means of a Survey Monkey questionnaire sent out to surgeons in NHS Grampian / Highlands and Tayside and a different Survey Monkey questionnaire sent to patients attending surgical outpatients in NHS Grampian.

SECONDARY OUTCOMES:
Are there any new surgical patients that can be seen or assessed by video or telephone consultation? Do remote consultations improve efficiency? | June 2021
  Analysis of the results of patient and surgeons' questionnaires will be undertaken to establish whether there are any types of new surgical patients that need not be seen face to face prior to the day of operation.
  Analysis of results from patient and surgeons' surveys will be undertaken to establish which type of surgical consultation (video, telephone or remote) is most appropriate in different clinical circumstances and this will be fed back to surgical outpatient department to assess impact on outpatient administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No